CLINICAL TRIAL: NCT03328962
Title: An Intervention Study of a Smoking Cessation Program Offered to Newly Diagnosed Cancer Patients at Their First Consultation for Treatment at an Oncological Hospital Department
Brief Title: Smoking Cessation in Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Norwegian Cancer Society (Other); Helse Stavanger HF (Other Government); Oslo University Hospital (Other); Sorlandet Hospital HF (Other Government); University Hospital of North Norway (Other); Helse Møre og Romsdal HF (Other Government); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Arnfinn Helleve, Researcher, Norwegian Institute of Public Health
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NorwegianIPH-001
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Smoking Cessation; Motivation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: The intervention group will receive structured smoking cessation counselling based on MI and adapted for the cancer setting combined with provision of smoking cessation medication (nicotine replacement therapy) while in the control group there will be standard care which may vary from hospital to hospital (intervention program and standard care will be described in details later).
  The recruitment period for the control group will be from September 2017 to March 2018. Participants in the control group will be invited to answer a follow up questionnaire after 6 months. Six months after the last recruited participant to the control group, i.e. from September 2018, recruitment of participants to the intervention group will begin and last for six months, to the end of February 2019 and the participants in the intervention group will be followed for 6 months, to the end of August 2019. The figure below gives an overview of the timing of recruitment and observations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Newly diagnosed cancer patients at their first consultation for treatment at an oncological hospital Department, who report to be smoking, recruited from 15/09/17 to 15/3/18. Their smoking status will be observed over a period of six months.
- Intervention group (Experimental): Newly diagnosed cancer patients at their first consultation for treatment at an oncological hospital Department, who report to be smoking, recruited from 15/09/18 to 15/3/19. The intervention group will receive structured smoking cessation counselling based on MI and adapted for the cancer setting combined with provision of smoking cessation medication (nicotine replacement therapy) while in the control group there will be standard care which may vary from hospital to hospital. Their smoking status will be observed over a period of six months.
  Interventions: Behavioral: Structured smoking cessation counselling based on motivational interviewing (MI) and adapted for the cancer setting eventually combined with provision of smoking cessation medication

INTERVENTIONS:
Behavioral: Structured smoking cessation counselling based on motivational interviewing (MI) and adapted for the cancer setting eventually combined with provision of smoking cessation medication — structured smoking cessation counselling based on MI and adapted for the cancer setting eventually combined with provision of smoking cessation medication
  Arms: Intervention group

SUMMARY:
The intervention to be studied is a smoking cessation program offered to newly diagnosed cancer patients at their first consultation for treatment at an oncological hospital department.

DETAILED DESCRIPTION:
The theoretical basis for the smoking cessation program is motivational interviewing (MI), an established counselling method previously used in smoking cessation programs as well as in other behaviour change programs. MI is defined as "a directive, client-centred counseling style for eliciting behaviour change by helping clients to explore and resolve ambivalence" (Miller 1983, cited in a Cochrane report by Lindson-Hawley, N et al., 2015). The 2015 Cochrane review concluded that MI may help people to quit smoking, but underlined at the same time that there were huge variations in study quality and intervention implementations. To our knowledge, a MI-based smoking cessation program has to a very limited extent been tried in a hospital setting before.

The program includes a cessation kit with a few samples of different smoking cessation drugs (nicotine replacement therapy) and consists of at least four individual counselling sessions (30-60 min) and follow up as needed during six months with a trained smoking cessation counsellor. Counselling will take place at the hospital premises, in conjunction with scheduled cancer treatment sessions for the patients.

In the current study, two nurses or radiation therapists at each of the included hospitals will receive training in using MI in smoking cessation counselling. The Norwegian Directorate of Health's standard smoking cessation program based on MI will be modified to be appropriate for cancer patients in treatment. The Norwegian Cancer Society (NCS) will be responsible for the training and the adaptation of the program. NCS will cover on average a 50 percent position designated smoking cessation counselling at each cancer ward. Counselling (one to one counselling) will take place in connection with cancer treatment appointments, before or after (preferably before as patients might feel unwell or nauseas after treatment), except for the first appointment that will happen before cancer treatment starts. Each counselling session will last for approximately 30-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cancer patients
* Offered radiation, chemo or immuno therapy in a designated hospitals
* Current smokers or recent quitters (within the last six weeks)
* 18 years or older

Exclusion Criteria:

* Survival prognosis less than 12 months
* Suffering dementia or other mental illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Smoking status | After 6 months
  Daily, occasional or no smoking

CONTACTS AND LOCATIONS:
Locations (6):
- Norway (6):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordlandssykehuset, Bodø
  - Sørlandet Hospital, Kristiansand
  - Oslo University Hospital, Oslo
  - St. Olavs Hospital, Trondheim